CLINICAL TRIAL: NCT05753137
Title: Acupuncture as Adjuvant Therapy for Glaucoma - Protocol for a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CMUH111-REC3-210
Record Dates: First submitted 2023-01-29; First posted 2023-03-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma; Acupuncture; Intraocular Pressure
Keywords: Glaucoma; Acupuncture
MeSH Terms: conditions — Glaucoma | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ophthalmic Acupoint Treatment Group (Experimental): Ophthalmic acupoint treatment group will receive a total of 6 courses of treatment, once a week, a total of six weeks, 20 minutes each time.
  Acupuncture points: Fengchi(GB20), Cuanzhu(BL2), Sibai(ST2), Taiyang(EX-HN5), Hegu(LI4), Taichong(LR3), a total of six acupoints.
  Interventions: Other: Acupuncture
- Non-ophthalmological Acupoint Control Group (Placebo Comparator): Non-ophthalmological acupoint control group will receive a total of 6 courses of treatment, once a week, a total of six weeks, 20 minutes each time.
  Acupuncture points: Yinlingquan(SP9), Liangqiu (ST34),Xiajuxu(ST39), Yanglingquan (GB34), Shousanli(LI10), Sanyangluo(TE8), a total of six acupoints. The Non-ophthalmological acupoint control group points are not indicated for the treatment of ophthalmological related pathologies, and are not reported to improve ophthalmological function.
  Interventions: Other: Acupuncture placebo

INTERVENTIONS:
Other: Acupuncture — The treatment will take place once a week, over six weeks. The needles will placed in the body for 20 minutes. A total of 12 Needles(6 acupoints, bilaterally) will be used in each session.Participants in the treatment group will undergo acupuncture targeting ophthalmology-related acupuncture points, aiming to elicit the 'De Qi' sensation.
  Arms: Ophthalmic Acupoint Treatment Group
Other: Acupuncture placebo — A total of 12 Needles(6 acupoints, bilaterally) will be used in each session. Acupuncture points are different from the experimental group.The control group will receive minimum acupuncture stimulation targeting non-ophthalmic acupuncture points without the intention of achieving the 'De Qi' sensation.
  Arms: Non-ophthalmological Acupoint Control Group

SUMMARY:
This clinical trial used acupuncture as an adjunctive treatment for glaucoma patients. A randomized, controlled trial involving 50 subjects will be conducted and observed for 12 weeks to evaluate the clinical efficacy of acupuncture. This study aims to provide a reference for future clinical treatment guidelines.

DETAILED DESCRIPTION:
This clinical trial utilized acupuncture as an adjunctive treatment for glaucoma patients. It is estimated a randomized clinical trial that 50 subjects will be enrolled and observed for 12 weeks to evaluate the clinical efficacy of acupuncture, providing a reference for future clinical treatment guidelines. Participants will be randomly divided into two groups: Ophthalmic Acupoint Treatment Group and Non-ophthalmological Acupoint Control Group. Participants in the treatment group will undergo acupuncture targeting ophthalmology-related acupuncture points, aiming to elicit the 'De Qi' sensation. Conversely, the control group will receive minimum acupuncture stimulation targeting non-ophthalmic acupuncture points without the intention of achieving the 'De Qi' sensation. Both groups will undergo acupuncture therapy once a week for a total of six sessions and will be observed for twelve weeks. On each visit, intraocular pressure, blood pressure, and heart rate will be assessed. Questionnaires of Glaucoma Symptom Scale (GSS) and The Glaucoma Quality of Life-15 (GQL-15) will be performed. The data of central corneal thickness, optical coherence tomography angiography, optical coherence tomography, visual field, and best-corrected visual acuity will be collected and analyzed before acupuncture and in the 12th week.

ELIGIBILITY:
Inclusion Criteria:

1. Primary open angle glaucoma diagnosed at least 3 months ago.
2. Diagnosed with mild or moderate open angel glaucoma.
3. Use 1 or 2 kinds of glaucoma drugs.
4. Age ≥ 20 years old.
5. Participants sign the informed consent and cooperate with the experimental procedures.

Exclusion Criteria:

1. Accept any ophthalmic laser or surgery within one year.
2. High myopia.
3. Use of any drugs that affect intraocular pressure.
4. Visual acuity with correction lower than 0.2.
5. Previous or existing uveitis or retinopathy.
6. Unable to receive acupuncture treatment continuously or allergic to acupuncture needles.
7. Pregnancy or breastfeeding.
8. Refusal to sign the informed consent form.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-06-27 (Estimated); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure-pre-treatment | Every weeks pre-acupuncture treatment up to six weeks.
  Intraocular pressure (IOP) is the fluid pressure of the eye.TOPCON CT-80 Computerized Tonometer is used for measurement.The unit of value is mmHg.
Intraocular pressure-after-treatment | Every weeks 15 minutes after acupuncture treatment up to six weeks.
  Intraocular pressure (IOP) is the fluid pressure of the eye.TOPCON CT-80 Computerized Tonometer is used for measurement.The unit of value is mmHg.
Intraocular pressure-Change | Change from baseline intraocular pressure at 12 weeks.
  Intraocular pressure (IOP) is the fluid pressure of the eye. Tonometer is used for measurement.The unit of value is mmHg.

SECONDARY OUTCOMES:
Optical coherence tomography-RNFL symmety | Change from baseline RNFL symmety at 12 weeks.
  The optic disk and the RNFL are the principal sites of apparent glaucomatous damage which precedes glaucomatous visual field alterations. RNFL symmety and Retinal nerve fiber layer (RNFL) thickness measurements obtained with Optical coherence tomography employs low-coherence interferometry.The unit of value is %.
Optical coherence tomography-C/D ratio | Change from baseline C/D ratio at 12 weeks.
  The optic disk and the RNFL are the principal sites of apparent glaucomatous damage which precedes glaucomatous visual field alterations. The cup/disc (C/D) ratio as a standardised method to evaluate the optic nerve obtained with Optical coherence tomography employs low-coherence interferometry.
Optical coherence tomography angiography-RPC density | Change from baseline RPC density at 6 weeks.
  Optical coherence tomography angiography is a relatively new, non-invasive, dye-free imaging modality that provides a qualitative and quantitative assessment of the vasculature in the retina and optic nerve head. We use OCTA to complement visual field and OCT examinations to diagnose glaucoma, detect progression and evaluate the treatment of acupuncture. Using OCT angiograms, the RPC density was evaluated quantitatively. The unit of value is %.
Central corneal thickness | On the first and 12th week for baseline and follow up tracing.
  To measure mean values of central corneal thickness (CCT) obtained by specular microscopy.
Glaucoma Symptom Scale | On the first and 12th week for baseline and follow up tracing.
  The Glaucoma Symptom Scale (GSS) is a simple and brief glaucoma-specific questionnaire aimed at quantifying complaints and functional impairment in patients with glaucoma. We used 1998 version of the Glaucoma Symptom Scale (GSS; Lee et al., 1998) Questionnaire.The items include 10 ocular complaints, for each eye, a 5-level score is generated, ranging from 0 (complaint present and very bothersome) to 4 (complaint absent). This score is then transformed to a 0 to 100 scale, with 0 representing presence of a very bothersome problem and 100 representing absence of a problem.
Glaucoma Quality of Life - 15 | On the first and 12th week for baseline and follow up tracing.
  The GQL-15 questionnaire is composed of 15 items. A 5-point rating scale for the level of difﬁculty of each task totals a score from 0 to 75. A higher score signiﬁes a poorer .
Blood pressure | we measure blood pressure every weeks before and after acupuncture treatment of totally six weeks, and first and 12th week for baseline and follow up tracing.
  We measure the blood pressure of patient before and after acupuncture treatment .Both systolic and diastolic blood pressure will be measured.
Heart rate | we measure heart rate every weeks before and after acupuncture treatment of totally six weeks, and first and 12th week for baseline and follow up tracing.
  We measure the heart rate of patient before and after acupuncture treatment .
Best corrected visual acuity | Change from baseline best corrected visual acuity at 12 weeks.
  Best possible vision a an eye can see with corrective lenses, measured in terms of Snellen lines.
Visual field- mean deviation | Change from baseline visual field at 12 weeks.
  The visual field refers to the total area in which objects can be seen in the side (peripheral) vision as you focus your eyes on a central point. Visual field will measured with automated perimetry.The unit of value is dB.
Visual field- visual field index | Change from baseline visual field at 12 weeks.
  The visual field refers to the total area in which objects can be seen in the side (peripheral) vision as you focus your eyes on a central point. Visual field will measured with automated perimetry. Visual field index intuitive presentation may underestimate the visual loss.

CONTACTS AND LOCATIONS:
Overall Officials: LEE YU-CHEN, Ph.D, Study Director — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jonas JB, Aung T, Bourne RR, Bron AM, Ritch R, Panda-Jonas S. Glaucoma. Lancet. 2017 Nov 11;390(10108):2183-2193. doi: 10.1016/S0140-6736(17)31469-1. Epub 2017 May 31. PMID 28577860
- [Result] Quigley HA. Number of people with glaucoma worldwide. Br J Ophthalmol. 1996 May;80(5):389-93. doi: 10.1136/bjo.80.5.389. PMID 8695555
- [Result] Quigley HA, Vitale S. Models of open-angle glaucoma prevalence and incidence in the United States. Invest Ophthalmol Vis Sci. 1997 Jan;38(1):83-91. PMID 9008633
- [Derived] Liao YF, Lee YC, Lin HJ, Shao YC. Acupuncture as Adjuvant Therapy for Glaucoma: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 8;13:e57888. doi: 10.2196/57888. PMID 39378079